CLINICAL TRIAL: NCT02043028
Title: Kneeling Posture With a Kneeling Stool During Cardiopulmonary Resuscitation in Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Jaehoon Oh, Department of Emergency Medicine, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Kneeling Posture; University of Ulsan 2013-0141 (Other Grant/Funding Number: University of Ulsan 2013-0141)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cardiac Arrest
Keywords: Cardiopulmonary resuscitation; Chest compression; Advanced cardiac life support; Posture
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Participants compress the chest of a manikin with kneeling posture using a kneeling stool for chest compression posture during 5 minutes
  2 weeks later, They perform the chest compression with standing posture using a step stool during 5 minutes
  Interventions: Device: Chest compression with a step stool; Device: Chest compression with a kneeling stool
- Group 2 (Experimental): Participants compress the chest of a manikin with a standing posture using a step stool for chest compression posture during 5 minutes
  2 weeks later, They perform the chest compression with a kneeling posture using a kneeling stool stool and bed height adjustment during 5 minutes
  Interventions: Device: Chest compression with a step stool; Device: Chest compression with a kneeling stool

INTERVENTIONS:
Device: Chest compression with a step stool — Participants compress the chest of a manikin with a standing posture using a step stool during 5 minutes
Device: Chest compression with a kneeling stool — Participants compress the chest of a manikin with kneeling posture using a kneeling stool during 5 minutes

SUMMARY:
To perform chest compression (CC) in the kneeling posture in hospital, we designed a stage with stairs, named the 'kneeling stool', on which a CC performer kneels beside a patient on a bed.This work is the validation study to demonstrate that the kneeling stool could be used for high quality hospital cardiopulmonary resuscitation (CPR) with the kneeling posture. We hypothesized that the quality of chest compression with a kneeling posture using the kneeling stool is equal to or superior to CC with a standing posture using the height adjustment mechanism of the bed.

DETAILED DESCRIPTION:
We designed and implemented the kneeling stool to perform CPR with the kneeling posture for a patient on a bed. The frame is constructed of an aluminum alloy. The size is 570 mm (width) x 598 mm (depth) x 600 mm (height). The weight is 9.3 kg, which is easily moved as needed. For easy rotation between rescuers, a step plate was inserted. To prevent pain to the knees of the kneeling CC performer, a 40mmthick sponge cushion was placed on the top plate and fixed to the frame.

A standard hospital bed frame (Transport stretcher®, 760 x2110 mm, 228 kg, Stryker Co., Kalamazoo, Michigan, USA), a foam mattress (660 x 920 x 80 mm, soft foam with polyurethane coverage, Stryker Co., USA), a backboard (450 ×600 ×10 mm, 3 kg Lifeline Plastic, Sung Shim Medical Co., Bucheon, Korea), and a step stool (395 x 450 x 410 mm, Gunica Co., Gyeongsangnam-do, Korea) were used in the experiment. A Resusci Annie Modular System Skill Reporter® manikin (Laerdal Medical, Orpington, UK) was used to perform CPR in the evaluations. We added weight to the manikin to equal 34 kg for simulating the upper body weight of an adult human as in a previous study.

Data collection The participants were divided into two groups by random drawing. Each performer in the first group knelt on the kneeling stool beside the manikin on a bed and compressed the chest of the manikin (CCs with a kneeling posture, PK).Each performer in the second group stood on a step stool beside the manikin on a bed and compressed the chest of the manikin (CCs with a standing posture, PS). When the performer stood beside the manikin on a bed, the height of the manikin's back was adjusted in height to the knee level of the provider using the step stool and the bed height adjustment mechanism. All the participants performed continuous CCs for 5 minutes without audio-visual feedback. After 2 weeks, the posture used for the CCs by each group was changed. Each participant recorded his/her fatigue and pain levels on a visual analogue scale (VAS, score 0 indicates "no pain and fatigue" and score 10 indicates "unbearable pain and fatigue") for each minute during 5 minutes of CCs. After conclusion of the experiment, the participants selected a preferred CC posture in terms of the safety and the quality of the CCs.

ELIGIBILITY:
Inclusion Criteria:

* Doctors and nurses working at emergency department
* American Heart Association Basic Life Support (AHA BLS) provider certification

Exclusion Criteria:

* Heart, wrist, or low back disease or who were pregnant were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Chest compression parameter | one day
  Chest compression depth and rate Accuracy of chest compression depth at least 5cm Incomplete chest recoil

SECONDARY OUTCOMES:
Visual analog scale(VAS) score of the overall fatigue and pain during chest compression | one day
  the VAS score ( 0, no fatigue pain to 10, unbearable) for the fatigue and pain during and after chest compression.

CONTACTS AND LOCATIONS:
Overall Officials: Jaehoon Oh, M.D., Principal Investigator — Department of emergency medicine, college of medicine, Hanyang university
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea